CLINICAL TRIAL: NCT03978013
Title: Pomegranate Juice Effect on Oxidative Stress in Infertile Women During IVF Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ola Gutzeit MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 017319
Record Dates: First submitted 2019-06-02; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: PCOS; Endometriosis; Advised Maternal Age; Male Factor Infertility
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pomegranate and control juice will be provided by Primor Company, Hadera, Israel. Control juice has similar color and test but do not include pomegranate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate (Experimental)
  Interventions: Other: Pomegranate juice
- Apple (Active Comparator)
  Interventions: Other: Apple juice

INTERVENTIONS:
Other: Pomegranate juice — Pomegranate juice
  Arms: Pomegranate
Other: Apple juice — Apple juice
  Arms: Apple

SUMMARY:
tTe investigators estimate pomegranate supplementation effect on oxidative stress in infertile women with PCOS, endometriosis and advanced maternal age during IVF treatment. The primary aim is to compare the obtained oxidative stress markers in follicular fluid with pomegranate supplementation vs control.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo IVF treatment with diagnosis of PCOS/Endometriosis/MF or AMA

Exclusion Criteria:

* Patients who do not meet the inclusion criteria, as above

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Cytokines levels in follicle fluid | 2 weeks
  Cytokines (pg/mL) will be mesured by elisa.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code